CLINICAL TRIAL: NCT00952081
Title: A Pilot Study to Evaluate Efficacy and Safety of Clevidipine in Neurosurgical Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-745
Record Dates: First submitted 2009-07-29; First posted 2009-08-04 (Estimated); Results first posted 2013-10-30 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: Hypertension; Brain Tumor; Epilepsy
Keywords: Hypertension; Neurosurgery; bloodpressure control; brain tumor resection; epilepsy focus resection
MeSH Terms: conditions — Hypertension; Brain Neoplasms; Epilepsy | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- clevidipine,brain tumor,hypertension (Experimental): 21 or older, Clevidipine in brain tumor resection, epilepsy focus resection during acute hypertension under general anesthesia
  Interventions: Drug: Clevidipine

INTERVENTIONS:
Drug: Clevidipine — Clevidipine (0.5 mg/ml in 20 % lipid solution) will be administered via peripheral vein using syringe pump; drug infusion will be initiated at 5 mg/hr (10ml/h) and titrated to effect up to a maximum rate of 32 mg/hr when SBP exceeds 130 mm Hg. The anesthesiologist will be allowed to administer the alternative antihypertensive treatment (e.g. labetalol, hydralazine) after achieving a maximum clevidipine infusion rate.
  Other Names: Cleviprex; Clevidipine butyrate

SUMMARY:
This protocol describes a study to gain experience in the use of Clevidipine for perioperative blood pressure control in patients undergoing craniotomy for brain tumor or epilepsy focus resection. The purpose of this study is to establish the efficacy of Clevidipine for intraoperative blood pressure control in patients undergoing intracranial procedures, and gather information on the dosage and adverse effects of Clevidipine in neurosurgical patients. This initial pilot experience serves to familiarize the investigators with the use of this drug prior to initiating a planned randomized trial versus institutional standard-of-care therapy. The investigators will obtain greater familiarity with the dosing of clevidipine in this patient population and collect information on the incidence of adverse effects.

DETAILED DESCRIPTION:
Clevidipine, a recently introduced, short-acting, vascular-selective calcium antagonist, could be a potentially useful adjuvant for neurosurgical cases. It decreases arterial blood pressure by reducing systemic vascular resistance with no effect on venous capacitance vessels (7). Clevidipine was successfully used for the treatment of hypertension in cardiac surgical patients (8). However, there is no information available on its efficacy and safety in patients undergoing intracranial surgery.

The perioperative course of patients undergoing intracranial surgery is frequently complicated by acute hypertensive episodes. Acute hypertension in neurosurgical patients is associated with intracranial bleeds and prolonged hospital stay (1). Even with current neuroanesthesia management, hemodynamic stability may be challenging, especially in hypertensive patients. An anesthetic technique that improves perioperative hemodynamics without increasing the incidence of undesirable events (such as increased intracranial pressure, prolonged recovery, etc.) is desirable.

A number of antihypertensive agents are available to treat perioperative hypertension. Labetalol is commonly used to treat hypertensive episodes in patients undergoing craniotomy, but may not be desirable in certain patient populations because of its low potency, a slow onset of peak effect (2), and unpredictability in dose requirements (3). Esmolol is only mildly effective in treating postoperative hypertension. Perioperative use is further complicated by bradycardia and conduction delay. Nicardipine is more effective than esmolol in controlling postoperative hypertension (4). However, it causes a dose-dependent cerebral vasodilation, inhibition of autoregulation, as well as a high incidence of hypotension (as compared to labetalol) (5). Hydralazine may increase intracranial pressure by as much as 100% and is rarely used as the sole agent in treating hypertension in neurosurgical patients (6).

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Able to give consent
* No significant laboratory abnormalities
* Undergoing elective surgery for tumor resection or epilepsy focus resection

Exclusion Criteria:

* Patients with acute cardiac ischemia, renal or liver dysfunction, unstable hemodynamic, advanced heart block, or pregnancy defective lipid metabolism such as pathologic hyperlipemia, lipoid nephrosis, or acute pancreatitis if it is accompanied by hyperlipidemia; and in patients with severe aortic stenosis will be excluded.
* Known or suspected allergy to study drug or study drug components,patients with allergies to soybeans, soy products, eggs, or egg products; Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Bekker, MD, PhD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, Department of Anesthesiology, New York, New York, United States

REFERENCES:
- See also: pubmed abstract — http://www.ncbi.nlm.nih.gov/pubmed/20622687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for intracranial surgery were prospectively enrolled after giving consent. Clevidipine (0.5 mg/mL in 20% lipid solution, which was to be initiated at 10 mg/h and titrated to effect) was administered as the primary antihypertensive agent for perioperative hypertension, with target BPs of less than 130mm Hg.
Groups:
- Clevidipine,Brain Tumor,Hypertension: Clevidipine(0.5 mg/mL in 20% lipid solution), initiated at 10 mg/h and titrated to effect, was administered as the primary antihypertensive agent for perioperative hypertension, with target BPs of less than 130mm Hg.
Period: Overall Study
Arm/Group | Clevidipine,Brain Tumor,Hypertension
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clevidipine,Brain Tumor,Hypertension
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (14.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of This Trial is the Proportion of Patients Who Did Not Require Rescue Antihypertensive Medication to Maintain SBP Below 130 mmHg (i.e. Clevidipine is a Sole Antihypertensive Agent Used for Blood Pressure Control)
Time Frame: intraoperatively and 90 min after surgery
Measure: Number; unit: participants
Arm/Group | Clevidipine,Brain Tumor,Hypertension
Number analyzed (Participants) | 22
participants | 21

ADVERSE EVENTS:
Description: Only Adverse Events attributed to study drug (clevidipine) were reported.
Arm/Group | Clevidipine,Brain Tumor,Hypertension
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No